CLINICAL TRIAL: NCT03191422
Title: LSVT BIG for Chronic Stroke Rehabilitation: a Single-Case Experimental Design
Brief Title: LSVT BIG for Chronic Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Valerie Metcalfe, Master's Candidate, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H03-16-07
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Chronic Stroke
Keywords: Rehabilitation; Occupational Performance

STUDY DESIGN:
Intervention Model Description: Single-Case experimental design One repetition
Masking Description: Outcome Assessor's for 2 of the outcome measures were blinded to the order of the pre and post assessment videos for rating, as well as being unfamiliar with the intervention protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LSVT BIG intervention recipients (Experimental): Participants participated in all of the evaluation steps as well as the LSVT BIG protocol which includes 16, 1-hour intervention sessions with a certified therapist performing, targeted exercises and activities to improve participation in occupations - with a focus on large amplitude movement.
  Interventions: Behavioral: LSVT BIG

INTERVENTIONS:
Behavioral: LSVT BIG — LSVT BIG is a motor learning based intervention 4 hour long sessions per week for 4 weeks following a specific protocol. Each session is composed of exercises and participant specific activities, as well as a homework program.

SUMMARY:
This study aims to explore if the LSVT BIG® - a motor learning based treatment program designed for rehabilitation of people with Parkinson's disease could be beneficial for chronic stroke rehabilitation. A single-case experimental design with two adult participants, will be monitored for performance on self-selected goals before, during and after participating in the treatment program.

DETAILED DESCRIPTION:
Over 700 000 Canadians are living with the effects of stroke. Approximately 60% of people living with the effects of stroke need help with every day activities and 84% are limited in the activities which they would like to participate in. Much research has focused on interventions for acute and sub-acute rehabilitation but it is also known that gains can still be made in the chronic stage. Among common rehabilitation interventions to reduce impairment, there is moderate evidence of effectiveness of constraint induced movement therapy (CIMT) and mirror therapy and weak evidence of effectiveness of repetitive task training. However, positive effects on impairment do not necessarily carryover into activities of daily living.

Therefore, an intervention program with a goal of improvement in occupational performance outside of the clinical setting, one that targets everyday activities and participant selected activities, would be a valuable tool for occupational therapy post stroke. The objective of this study was to explore whether the LSVT BIG® program, an intervention targeting participant-identified functional goals which includes strategies to encourage generalization to other tasks, could be applicable to the rehabilitation of the chronic effects of stroke.

LSVT BIG is a time limited, high intensity rehabilitation program designed to be used by occupational therapists or physiotherapists to target Parkinson's disease motor symptoms of bradykinesia and hypokinesia, in an outpatient environment, with a goal of improving function. This intervention involves exercises and repetitive practice of patient-selected activities with a focus on big (increased amplitude) movements. It is believed that this will lead to normally paced and sized movements which will generalize to untrained activities.

Although Parkinson's disease and stroke have different pathological mechanisms, the elements in the LSVT BIG program are based on the same neuroplasticity and motor learning principles that form the basis for stroke rehabilitation methods. What is novel, however, is the focus on amplitude and just one cue, 'big', for all difficult movement situations, potentially increasing generalizability outside of the clinical setting and trained activities.

The LSVT BIG program uses motor learning principles of blocked practice, serial practice and elements of random practice (varying environmental factors), extrinsic feedback (including verbal feedback, modeling, shaping and focus on knowledge of results) as well as a single external, knowledge of results focused cue 'big' to encourage adaptation, recalibration of the internal motor program of the movement, and transfer to other tasks. LSVT BIG also respects the neuroplasticity principles of intensity, repetition, specificity and saliency The aim of this study is to begin to explore the effectiveness of LSVT BIG in late stroke rehabilitation.

The primary hypothesis is that participants with chronic stroke will demonstrate improvement in trained activities following LSVT BIG.

A secondary hypothesis is that participants will also improve in untrained activities due to carryover of the intervention effects.

Study Design A single-case experimental design (SCED) with one replication was used . An A-B-A design was selected and included a baseline phase, an intervention phase, and a post-intervention phase. Perceived performance and satisfaction with performance of participant-selected activities, and self-report of everyday upper extremity use were the outcomes subjected to repeated measures. In addition, pre- and post- measures of observed performance quality and upper extremity function were carried out.

ELIGIBILITY:
Inclusion Criteria:

* stroke at least 6 months previously,
* communication in english or french,
* adequate cognition to follow direction and complete independent homework,
* independent mobility,
* medical stability,
* minimum Stage 3 for arm and hand on the Cherokee McMaster Stroke Assessment

Exclusion Criteria:

* dementia,
* psychiatric disorder,
* medical condition that would prevent participation in aerobic exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Change in perceived occupational performance | Administered weekly, for 6 weeks pre-intervention, 4 weeks during intervention and 5 post-intervention
  Positive change on performance score using the Canadian Occupational Performance Measure (COPM)

SECONDARY OUTCOMES:
Perceived changes in upper extremity use | Administered weekly, for 6 weeks pre-intervention, 4 weeks during intervention and 5 post-intervention
  Positive change in perceived upper extremity use using the Rating of Everyday Arm-Use in the Community and Home (REACH)
Objective rating of activity performance | Administered at week 1 and week 10
  Positive change in objective rating of activity performance using the Performance Quality Rating Scale- Operational Definition (PQRS-OD),
Rating of upper extremity function | Administered at week 1 and week 10
  Positive change in upper extremity function as measured by the Chedoke Arm and Hand Activity Inventory-13(CAHAI-13)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Metcalfe, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share data.